CLINICAL TRIAL: NCT00130104
Title: Transthecal Metacarpal Block vs Traditional Digital Block for Painful Finger Procedures in Children
Brief Title: Transthecal Metacarpal Block Versus Traditional Digital Block for Painful Finger Procedures in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-5-4319
Record Dates: First submitted 2005-08-11; First posted 2005-08-15 (Estimated); Last update posted 2007-10-05 (Estimated); Status verified 2005-08

CONDITIONS: Finger Injuries
Keywords: digital block; regional anesthesia; finger repair; Fingers; Anesthesia, Conduction
MeSH Terms: conditions — Finger Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- MCB (Experimental): randomized to receive the metacarpal block for anesthesia
  Interventions: Procedure: Transthecal Metacarpal Block

INTERVENTIONS:
Procedure: Transthecal Metacarpal Block

SUMMARY:
The purpose of this study is to determine if the transthecal metacarpal block is superior to the traditional digital block for regional digital anesthesia in children.

DETAILED DESCRIPTION:
Background: Finger injuries and infections are common presenting problems in the pediatric emergency department. A traditional digital block, requiring at least two injections of anesthetic, is the traditional method of regional anesthesia for many finger procedures. Digital blocks can sometimes be difficult to administer and assess for effectiveness especially in children. A newer procedure, the transthecal metacarpal block, may be easier to administer, and more effective with one injection.

Objective: To determine if the transthecal metacarpal block (MCB) provides superior digit anesthesia in children requiring painful finger procedures as compared to the traditional digital block (TDB).

Methods: A randomized clinical trial comparing the MCB to the TDB will be conducted in an urban, tertiary care pediatric emergency department. Children <18 years of age, presenting to the emergency department with a finger injury or infection, which requires regional anesthesia for repair will be screened for eligibility. Eligible patients, with appropriate consent will be randomized to receive either the MCB or TDB with 1% Lidocaine. The primary outcome, success of the block will be assessed using pinprick testing after a standardized wait time. Secondary outcomes including pain with the block and repair, repairing physician satisfaction, and short-term complications will also be assessed.

Implications: Finding successful methods of anesthesia and pain control are paramount in the pediatric emergency department. In addition, using a type of digital block which is easy to administer, successful, and requires only one injection would give physicians confidence to treat finger injuries in children with regional anesthesia and possibly avoid procedural sedation in some cases. To date, no studies have been published on the efficacy of digital blocks in children. This study will also serve to give baseline success rates for both types of digital blocks.

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years
* Greater than 10 kg in weight
* Have finger injuries or infections that will require digital regional anesthesia
* Require only local anesthesia for the repair
* English speaking

Exclusion Criteria:

* Have previous participation in this study
* Need procedural sedation at the onset of the repair
* Have allergy to lidocaine or amide-type local anesthetics
* Have infection at the sites of block injection
* Have known coagulopathy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2005-07; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Success of the two types of digital blocks | immediate

SECONDARY OUTCOMES:
Pain experienced with the digital block | immediate
Repairing physician satisfaction with the procedure | immediate
complications associated with digital block | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Alpern, MD, MSCE, Principal Investigator — The Children's Hospital of Philadelphia, Division of Emergency Medicine
Locations (1):
- The Children's Hospital Of Philadelphia Emergency Department, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Bhende MS, Dandrea LA, Davis HW. Hand injuries in children presenting to a pediatric emergency department. Ann Emerg Med. 1993 Oct;22(10):1519-23. doi: 10.1016/s0196-0644(05)81251-x. PMID 8214828
- [Background] Kelly JJ, Spektor M. Nerve Blocks of the Thorax and Extremities. In:Roberts J, Hedges J, eds. Clinical Procedures in Emergency Medicine. St. Louis: WB Saunders, 2004.
- [Background] Robson AK, Bloom PA. Suturing of digital lacerations: digital block or local infiltration? Ann R Coll Surg Engl. 1990 Nov;72(6):360-1. PMID 2241053
- [Background] Flarity-Reed K. Methods of digital block. J Emerg Nurs. 2002 Aug;28(4):351-4. doi: 10.1067/men.2002.125539. No abstract available. PMID 12122413
- [Background] Chiu DT. Transthecal digital block: flexor tendon sheath used for anesthetic infusion. J Hand Surg Am. 1990 May;15(3):471-7. doi: 10.1016/0363-5023(90)90063-w. PMID 2348068
- [Background] Brutus JP, Baeten Y, Chahidi N, Kinnen L, Ledoux P, Moermans JP. Single injection digital block: comparison between three techniques. Chir Main. 2002 May;21(3):182-7. doi: 10.1016/s1297-3203(02)00107-5. PMID 12116830
- [Background] Cummings AJ, Tisol WB, Meyer LE. Modified transthecal digital block versus traditional digital block for anesthesia of the finger. J Hand Surg Am. 2004 Jan;29(1):44-8. doi: 10.1016/j.jhsa.2003.09.018. PMID 14751102
- [Background] Low CK, Vartany A, Engstrom JW, Poncelet A, Diao E. Comparison of transthecal and subcutaneous single-injection digital block techniques. J Hand Surg Am. 1997 Sep;22(5):901-5. doi: 10.1016/S0363-5023(97)80088-3. PMID 9330152
- [Background] Morrison WG. Transthecal digital block. Arch Emerg Med. 1993 Mar;10(1):35-8. doi: 10.1136/emj.10.1.35. PMID 8452611
- [Background] Torok PJ, Flinn SD, Shin AY. Transthecal digital block at the proximal phalanx. J Hand Surg Br. 2001 Feb;26(1):69-71. doi: 10.1054/jhsb.2000.0519. PMID 11162023
- [Background] Hill RG Jr, Patterson JW, Parker JC, Bauer J, Wright E, Heller MB. Comparison of transthecal digital block and traditional digital block for anesthesia of the finger. Ann Emerg Med. 1995 May;25(5):604-7. doi: 10.1016/s0196-0644(95)70171-0. PMID 7741335
- [Background] Hollander JE, Valentine SM, Brogan GX Jr. Academic associate program: integrating clinical emergency medicine research with undergraduate education. Acad Emerg Med. 1997 Mar;4(3):225-30. doi: 10.1111/j.1553-2712.1997.tb03747.x. PMID 9063553
- [Background] Castellanos J, Ramirez C, De Sena L, Bertran C. Transthecal digital block: digital anaesthesia through the sheath of the flexor tendon. J Bone Joint Surg Br. 2000 Aug;82(6):889. doi: 10.1302/0301-620x.82b6.10430. PMID 10990318
- [Background] Lewis L, Stephan M. Local and Regional Anesthesia. In: Henretig F, King C, eds. Pediatric Emergency Procedures. Baltimore: Williams and Wilkins, 1997.
- [Background] Carlson D, et al. Illustrated Techniques of Pediatric Emergency Procedures. In: Fleisher G, Ludwig S, eds. Pediatric Emergency Medicine. Philadelphia: Williams and Wilkins, 2000.
- [Background] Antevy PM, Zuckerbraun NS, Saladino RA, Pitetti RD. Evaluation of a transthecal digital nerve block in the injured pediatric patient. Pediatr Emerg Care. 2010 Mar;26(3):177-80. doi: 10.1097/PEC.0b013e3181d1dfaf. PMID 20179662